CLINICAL TRIAL: NCT01545544
Title: Observational Study of B-Cell Non Hodgkin Lymphomas (NHL) in Patients With Hepatitis C Virus
Brief Title: Observational Study of B-Cell Non Hodgkin Lymphomas (NHL) Associated With Hepatitis C Virus (HCV)
Acronym: Lympho C
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS HC13 Lympho C
Record Dates: First submitted 2012-02-21; First posted 2012-03-06 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Hepatitis C
Keywords: B-Cell Non Hodgkin Lymphomas; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — whole blood and bone marrow
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An prospective / retrospective multicenter observational study whose objectives are to understand the interactions between hepatitis c virus and Non Hodgkin lymphomas. The characteristics , evolution and treatment of diseases will be observed from the study.

DETAILED DESCRIPTION:
Main objectives are:

* Description of the clinical and histological characteristics, treatment and evolution of these NHL.
* Study their physiopathology by immunological, virologic and molecular studies.

The study included prospective or retrospective patients with B- Cell Non-Hodgkin lymphomas (NHL) associated with chronic hepatitis C. The patients are diagnosed or in remission of lymphoma, in relapse or failure of treatments.

The enrolment period is 6 years and the total study lasts 8 years.

* "Prospective patients" are followed every 6 months during one year, and all the years during 2 or 5 years.
* "Retropective patients" are followed all the years during 2 or 5 years. At each follow-up, a blood sample of 50ml is withdrawn allowing ancillary studies.

The enrollment is estimated at 140 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evolving NHL whatever its histological type
* At diagnosis or relapse or failure previous treatments stopped over 3 months
* Patients with HCV infection with positive quantitative viral load
* 18 years or more of age
* Life expectancy greater than 6 months
* Signed and informed consent
* Benefit from social security

Exclusion Criteria:

* Active uncontrolled infection (out hepatitis C)
* HIV (Human immunodeficiency virus) infection
* Severe psychiatric history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HCV infection with positive viral load and a B-cell NHL.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2006-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
presentation of NHL and HCV infection, and treatments of NHL and HCV infection | at the first visit (Day 0)
  the presentation of NHL and HCV infection is done by clinical,histological and biological characteristics

SECONDARY OUTCOMES:
Summary of intercurrents biological and clinical events | Month 6, Month 12, Month 24, Month 36, Month 48 and Month 60
virological response | Month 60
  HCV quantitative viral load
haematological response | Month 60
  to evaluate the correlation between hematological and virological response

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HERMINE, PU-PH, Principal Investigator — Hôpital Necker (Paris 15è), Service d'hématologie; Fabrice CARRAT, PU-PH, Study Chair — Unité INSERM 707
Locations (1):
- Hôpital Necker, Paris, France

REFERENCES:
- [Derived] Michot JM, Canioni D, Driss H, Alric L, Cacoub P, Suarez F, Sibon D, Thieblemont C, Dupuis J, Terrier B, Feray C, Tilly H, Pol S, Leblond V, Settegrana C, Rabiega P, Barthe Y, Hendel-Chavez H, Nguyen-Khac F, Merle-Beral H, Berger F, Molina T, Charlotte F, Carrat F, Davi F, Hermine O, Besson C; ANRS HC-13 Lympho-C Study Group. Antiviral therapy is associated with a better survival in patients with hepatitis C virus and B-cell non-Hodgkin lymphomas, ANRS HC-13 lympho-C study. Am J Hematol. 2015 Mar;90(3):197-203. doi: 10.1002/ajh.23889. Epub 2014 Nov 24. PMID 25417909
- See also: Related Info — http://anrs.fr